CLINICAL TRIAL: NCT05561894
Title: Effects of Two Different Goals of Fluid Management in Patients Undergoing Supratentorial
Brief Title: Effects of Two Different Goals of Fluid Management in Patients Undergoing Supratentorial Tumour Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ibraheem Abdelmageed, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: master 1
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Supratentorial Brain Tumor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (control) (Placebo Comparator): Brain tumor excision under general anesthesia. Intervention (Pulse pressure variation index guided fluid therapy): PPVI will be measured using invasive blood pressure monitor. Ringer acetate solution will be administrated whenever PPV is higher than 12%.
  Interventions: Other: pulse pressure variation index guided fluid therapy
- B (Active Comparator): Brain tumor excision under general anesthesia. Intervention (Pulse pressure variation index guided fluid therapy): PPVI will be measured using invasive blood pressure monitor. Ringer acetate solution will be administrated whenever PPV is higher than 16%.
  Interventions: Other: pulse pressure variation index guided fluid therapy

INTERVENTIONS:
Other: pulse pressure variation index guided fluid therapy — maintainence intraoperative fluid therapy (ringer's acetate) will be given guided by either two goals of pulse pressure variation index, either >12% or >16%

SUMMARY:
Neurosurgical operations are characterised by major fluid shift, frequent use of diuretics, and prolonged operative time. The role of fluid therapy in these patients is very critical; hypovolemia might decrease cerebral perfusion; while, fluid over-infusion might swell the brain (1-3). Thus, fluid management in these procedures complex and challenging. Evidence on the optimum protocol for intraoperative fluid management in neurosurgical patients is still lacking. Adequate intracranial volume management is considered a key factor that would overcome the tumour bulk and the surrounding vasogenic oedema facilitating surgical access . Thus, a relaxed brain is one of the targets of intraoperative fluid management during craniotomy. The slack brain would allow proper surgical retraction and consequently, reduces brain retractor ischemia. Brain relaxation scale (BRS) had shown a good correlation with intracranial pressure thus, an increasing interest was paid to BRS as a simple surrogate for intracranial pressure (4-8).

Goal-directed hemodynamic therapy (GDT) in the operating room is a term used to describe the use of defined hemodynamic targets to guide intravenous fluid and inotropic therapy. Pulse pressure variation (PPV) is one of the robust dynamic indices of fluid responsiveness which is based on heart-lung interactions (9-12). GDT had been frequently investigated in the operating room in high-risk patients especially in major surgery. However, the impact of GDT on patient outcomes, especially BRS, is not well evaluated in brain surgery (12-15). In this study, we evaluated PPV-guided fluid management compared to standard fluid management in patients undergoing supratentorial mass excision. We hypothesised that in these procedures, GDT might restrict intraoperative fluid volume, improve brain relaxation, and provide stable patient hemodynamics.

DETAILED DESCRIPTION:
Anesthetic management:

Peripheral i.v line will be inserted and 2-3 mg midazolam and 2 gm magnesium are given. A pre-induction radial arterial line is inserted with the aid of infiltration of 2 ml lidocaine 2%. Invasive arterial blood pressure monitoring is started and pulse oximetry, 5-leads ECG, and NIBP are attached to the patient and mindray ipm-12 monitor is used. Anesthetic induction started with propofol 1-2 mg/kg, lidocaine 1 mg/kg, cis-atracurium 0.2 mg/kg and fentanyl 1-2 microgram/kg. Intubation is done with cuffed endotracheal tube and tidal volume and respiratory rate are set to achieve end-tidal Co2 of 30-28 mmHg. Esophageal temperature probe and urinary catheter are put in place. Patients then will receive maintenance of anesthesia with isoflurane < 1 MAC, propofol 10-60 microgram/kg/min, dexmedetomidine loading 1 microgram/kg bolus in 10 minutes followed by 0.2-1 microgram/kg/hour and cis-atracurium 2-3 microgram/kg/minute. Patients will receive mannitol 20% 0.5-1 gm/kg and dexamethasone 8mg and paracetamol 1gm near the end of surgery. Patients will receive their fasting requirements of normal saline in the first 3 hours of surgery. Maintenance fluid used will be ringer acetate and will be given according to pulse pressure variation index (PPVI) that is derived from pulse contour analysis of invasive arterial blood pressure waveform. Patients are then divided into two groups of two different targets of PPVI. Group A will be given ringer acetate when PPVI is > 12% and group B will be given ringer acetate when PPVI is > 16%.

If hypotension occurred without change in PPVI targets, it will be treated with 10 mg ephedrine. Arterial blood gas samples will be collected at induction and at the end of surgery. After removal of cranial fixation pins, anesthesia is discontinued and reversal of muscle relaxant is done with atropine 0.5 mg and neostigmine 0.05 mg/kg then extubation is done and patient is transferred to the ICU.

ELIGIBILITY:
Inclusion Criteria:

ASA 1,2 patients undergoing supratentorial tumour resection Age > 18 years Supine position

Exclusion Criteria:

* ASA 3,4 patients and patients with GCS < 13
* Any other position rather than supine position
* AF or any significant arrhythmia
* Severe bradycardia that leads to low HR/RR ratio
* Severe tricuspid regurgitation or severe right ventricular dysfunction
* Patients with severe restrictive lung pathology and needing low tidal volumes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
intraoperative mean arterial blood pressure | before induction of anesthesia as a baseline, after induction and then every 15 minutes till the end of surgery
  measured by invasive arterial blood pressure through radial arterial line

SECONDARY OUTCOMES:
postoperative adverse cardiovascular outcomes | 24 hours postoperative
  incidence of hypotension < 25% of baseline blood pressure
intraoperative urine output | at the end of surgery
  total amount of urine output at the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No